CLINICAL TRIAL: NCT05645965
Title: Association of Obesity and Cardiovascular Outcomes in Patients With Implantable Cardioverter-defibrillator (ICD) : a Korean Nationwide Cohort Study
Brief Title: Association of Obesity and Cardiovascular Outcomes in Patients With Implantable Cardioverter-defibrillator (ICD)
Acronym: Paradox
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Kwang-No Lee, Professor, Ajou University School of Medicine
Other Study IDs: AJOUIRB-EXP-2021-398-5
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Implantable Defibrillator User; Arrhythmias, Cardiac; Obesity; Cardiovascular Morbidity
Keywords: implantable cardioverter-defibrillator (ICD); obesity paradox
MeSH Terms: conditions — Arrhythmias, Cardiac; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent implantable cardioverter-defibrillator (ICD) insertion during study period: Patients who underwent implantable cardioverter-defibrillator (ICD) insertion between January 2015 and December 2020
  Interventions: Device: ICD insertion

INTERVENTIONS:
Device: ICD insertion — Patients who underwent implantable cardioverter-defibrillator (ICD) insertion between January 2015 and December 2020
  Other Names: Implantable cardioverter-defibrillator insertion

SUMMARY:
In this study, the investigators evaluated the association between various measures of adiposity [BMI and waist circumference (WC)] and clinical outcomes in Asian patients who underwent Implantable Cardioverter-defibrillator (ICD) insertion, using a nationwide population based cohort.

DETAILED DESCRIPTION:
This retrospective nationwide cohort study used administrative claims data from the Korean National Health Insurance Service (NHIS) and the combined health check-up database of the National Health Insurance Corporation between 2013 and 2020.

The investigators included patients who underwent implantable cardioverter-defibrillator (ICD) insertion between January 2015 and December 2020. Patients aged <20 years, those who were already taken ICD insertion before 2015, and those with cancer were excluded from the analysis. The follow-up period was defined as the time from the index date (date of device procedure) to each outcome event, date of death, or end of the study period (December 31, 2020), whichever came first.

Patients' demographic data, comorbidities, concomitant medications, and income level were collected from the Korean NHIS database. The recent health check-up data from the index date was also ascertained, including height, weight, waist circumference, blood pressure, health surveys, and laboratory exam. Health survey included family history, smoking history, alcohol history, and the level of individual physical activity.

According to BMI following the World Health Organization recommendation for Asian population, study patients were categorized into 5 groups: underweight, <18.5 kg/m2; normal range, 18.5 to <23 kg/m2; overweight, 23 to <25 kg/m2; obese I, 25 to <30 kg/m2; and obese II, ≥30 kg/m2[4]. The investigators defined the proportion of medical use by calculating formula with the recuperation cost and the number of the visit to hospitals.

During the follow-up period, the investigators assessed 3 clinical outcomes, including all-cause death, cardiovascular hospitalization and the recurrence rate. Clinical outcomes were mainly defined by the the International Classification of Diseases, 10th revision (ICD-10). Patients were censored at the clinical outcomes or the end of the study period (December 31, 2020), whichever came first.

All categorical variables are presented as frequencies and percentages. Normally distributed data were presented as mean ± standard deviation, whereas nonparametric data are presented as median and interquartile range by BMI.

Cox proportional hazard regression analyses were performed to identify the association of BMI with the primary and secondary outcomes, calculating hazard ratio (HR) and 95% confidence interval (CI) and adjusting for the following potential confounders: sex, age, systolic blood pressure, fasting glucose level, total cholesterol level, alcohol consumption, smoking status, physical activity, household income, use of antihypertensive agents, use of statins, use of antiplatelet agents, previous history of MI, previous history of stroke, and index year. All analyses were conducted using R-statistics.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent implantable cardioverter-defibrillator (ICD) insertion between January 2015 and December 2020

Exclusion Criteria:

* Patients aged <20 years
* Patients already taken ICD insertion before 2015
* Patients with cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We included patients who underwent implantable cardioverter-defibrillator (ICD) insertion between January 2015 and December 2020. Patients aged <20 years, those who were already taken ICD insertion before 2015, and those with cancer were excluded from the analysis.
  The follow-up period was defined as the time from the index date (date of device procedure) to each outcome event, date of death, or end of the study period (December 31, 2020), whichever came first.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of Outcomes | 5 years
  Death + CV hospitalization + Fatal arrest event + Infective endocarditis

SECONDARY OUTCOMES:
Death | 5 years
  Mortality
CV hospitalization | 5 years
  Admission caused by Cardiovacular disease
Fatal arrest event | 5 years
  Event of cardiac arrest by ventricular tachycardia and fibrillation
Infective endocarditis | 5 years
  Diagnosed with infective endocarditis

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-No LEE, Study Chair — Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim MS, Kim WJ, Khera AV, Kim JY, Yon DK, Lee SW, Shin JI, Won HH. Association between adiposity and cardiovascular outcomes: an umbrella review and meta-analysis of observational and Mendelian randomization studies. Eur Heart J. 2021 Sep 7;42(34):3388-3403. doi: 10.1093/eurheartj/ehab454. PMID 34333589
- [Background] Echouffo-Tcheugui JB, Masoudi FA, Bao H, Curtis JP, Heidenreich PA, Fonarow GC. Body mass index and outcomes of cardiac resynchronization with implantable cardioverter-defibrillator therapy in older patients with heart failure. Eur J Heart Fail. 2019 Sep;21(9):1093-1102. doi: 10.1002/ejhf.1552. Epub 2019 Jul 29. PMID 31359595
- [Background] Samanta R, Narayan A, Pouliopoulos J, Kovoor P, Thiagalingam A. Influence of Body Mass Index on Recurrence of Ventricular Arrhythmia, Mortality in Defibrillator Recipients With Ischaemic Cardiomyopathy. Heart Lung Circ. 2020 Feb;29(2):254-261. doi: 10.1016/j.hlc.2018.12.018. Epub 2019 Jan 30. PMID 30922553